CLINICAL TRIAL: NCT00945360
Title: Aromatase Inhibitors for the Prevention of the Growth of Uterine Leiomyomas in Perimenopausal Women: A Pilot Study
Brief Title: Aromatase Inhibitors for Treatment of Uterine Leiomyomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Anwar Nassar, MD/Associate Professor, American University of Beirut Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OGY.AN.08
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Symptomatic or Large Uterine Fibroids
Keywords: Leiomyoma; perimenopause; aromatase inhibitor
MeSH Terms: conditions — Leiomyoma | interventions — Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aromatase inhibitors: Letrozole (Experimental): All consenting patients will be started on Letrozole at a dose of 2.5 mg/day for 8 weeks.
  Interventions: Drug: Letrozole (aromatase inhibitor)

INTERVENTIONS:
Drug: Letrozole (aromatase inhibitor) — Letrozole at a dose of 2.5 mg/day for 8 weeks.
  Other Names: Letrozole

SUMMARY:
Fibroids are benign tumors that might results in bleeding. Surgery is their definitive treatment. Some medical therapies have been tried for women who wish to preserve their uterus. Recent reports have demonstrated a role for a new category of drugs called aromatase inhibitor (such as Femara) in the treatment of fibroids. This study is conducted to assess the effect of Femara (letrozole) on the size of fibroids in women around menopause.

DETAILED DESCRIPTION:
Fibroids (leiomyomas) are benign tumors that originate in the musculature of the uterus. They are the most common cause for removal of the uterus in women. Surgery is the final definitive treatment of fibroids. However, surgery is relatively risky. Hence, a few medical therapies have been tried for women who wish to preserve their uterus. However, most of those therapies have side effects that prohibit their routine use. Recent reports have demonstrated a role for a new category of drugs called aromatase inhibitor ( such as Femara) in the treatment of fibroids. To the best of our knowledge, this drug has not been studied yet in the management of fibroid of the uterus apart from one case report.

The objective of the current study is to assess the effect of aromatase inhibitors, specifically Femara (letrozole) on the size of fibroids in women around menopause. We are hoping that by decreasing their size, we could avoid having patients undergo surgery. The data generated is invaluable in that sense.

ELIGIBILITY:
Inclusion Criteria:

1. Perimenopausal women (≥ 50 years) with symptomatic uterine leiomyomas (menometrorrhagia, pressure symptoms, urinary retention, pelvic pain) or those with large leiomyomas ≥ 7 cms

Exclusion Criteria:

1. Women <50 years of age
2. Postmenopausal women
3. Women with impaired renal function
4. Oral treatment with any type of estrogen or progesterone more recently than 1 month
5. History of venous thromboembolism
6. Any contraindication for Magnetic Resonance Imaging (MRI)

Ages: 50 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary end point of this study will be the baseline to end point percent difference in leiomyoma volume at 2 months and 6 months following treatment with Letrozole. | 2 months and 6 months following treatment

SECONDARY OUTCOMES:
Improvement in symptoms | 2 and 6 months following treatment
Need for a surgical intervention | 2 and 6 months following treatment
Improvement in the hemoglobin levels | 2 and 6 months following treatment
Development of side effects: hot flushes, nausea,vomiting, headache, thrombophlebitis | 2 and 6 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anwar H Nassar, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon